CLINICAL TRIAL: NCT03880279
Title: A Phase I/II Trial Investigating Safety and Efficacy of Autologous TAC T Cells Targeting CD19 in Relapsed or Refractory Large B-Cell Lymphoma
Brief Title: Autologous TAC T Cells Targeting CD19 in R/R Large B-Cell Lymphoma
Acronym: TACTIC-19
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Following a change in company governance, Triumvira terminated the study prior to enrolling any subjects due to a challenging competitive landscape.
Sponsor: Triumvira Immunologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAC01-CD19-01
Record Dates: First submitted 2019-03-13; First posted 2019-03-19 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Lymphoma, B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TAC01-CD19 (Experimental): TAC01-CD19, Autologous TAC (T cell antigen coupler) T cells, single infusion, multiple dosage levels.
  Interventions: Biological: TAC01-CD19

INTERVENTIONS:
Biological: TAC01-CD19 — Dose-escalating cohorts plus expansion groups

SUMMARY:
Phase I/II study to evaluate TAC01-CD19 in subjects with relapsed or refractory B-cell lymphomas. TAC technology is a novel way to genetically modify T cells and to redirect these T cells to target cancer antigens by co-opting the natural T cell receptor. The dose finding portion of this study will evaluate the safety and tolerability of increasing dose levels of TAC01-CD19 to identify a Maximal Tolerated Dose (MTD) or Recommended Phase II Dose (RP2D). The dose expansion portion of the study will further evaluate the safety, efficacy and pharmacokinetics of TAC01-CD19 at the RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD19+ Large B-Cell Lymphoma including Diffuse Large B-cell Lymphoma (DLBCL) not otherwise specified (including de novo and transformed lymphoma), Primary Mediastinal Large B-cell Lymphoma, High-Grade B-cell Lymphoma with MYC and BCL2 and/or BCL6 rearrangement per WHO 2016 classification.
* Relapsed or refractory disease after greater than 2 lines of therapy including anthracycline and anti-CD20 therapy and either having failed autologous stem cell transplant (ASCT) or being ineligible for ASCT.
* ECOG 0-1.
* Adequate organ function.

Exclusion Criteria:

* Prior treatment with any of the following: allogeneic bone marrow transplantation, gene therapy, adoptive cell transfer of any kind, including CAR T cells.
* Active central nervous system (CNS) lymphoma involvement.
* History or presence of clinically relevant CNS pathology.
* Active inflammatory neurological disorders, autoimmune disease, or infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | First 28 days after dosing
  Measurement of occurrence of study-defined DLTs
Incidence of adverse events (AEs) | Informed consent through 2 years after dosing
  Type, frequency, and severity of adverse events (AEs) and laboratory abnormalities

IPD SHARING:
Plan to Share IPD: No